CLINICAL TRIAL: NCT07312786
Title: Testing the Feasibility of a Virtual Application to Support Breast and Colorectal Cancer Survivors After Completing Primary Treatment
Brief Title: Testing the Feasibility of a Virtual Application to Support Breast and Colorectal Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Robin Urquhart, NSHealth Affiliate Scientist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 707168
Record Dates: First submitted 2025-11-24; First posted 2025-12-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Survivor; Colorectal Cancer Survivors
Keywords: Cancer Survivorship; SeamlessMD; Supported self-management; Survivorship app

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual self-management intervention (Experimental)
  Interventions: Behavioral: virtual self-management intervention

INTERVENTIONS:
Behavioral: virtual self-management intervention — The intervention is a supportive information and self-management tool housed on the SeamlessMD mobile app, created in collaboration with the SeamlessMD development program and informed by foundational research. The application will be used as an information hub and self-management/navigation tool alongside usual care, to address the physical, psychosocial, and practical needs of breast and colorectal cancer survivors. Note that the intervention will not seek to change or impact a survivor's follow-up care plan, as decided upon by the participant and their care team.

SUMMARY:
The goal of this study is to determine the feasibility of implementing a mobile health application for breast and colorectal cancer survivors following primary treatment. Developed in collaboration with Seamless MD, the intervention acts as an information hub, providing users with timely and evidence-based information related to follow-up care as well as health system/community-based resources and programs to meet their needs during this period of care. The goal of the intervention is to encourage open communication regarding survivorship expectations and provide survivors with appropriate information and support to meet their needs.

This study will:

1. Test the feasibility of implementing the virtual intervention at two cancer centres in Atlantic Canada (Nova Scotia and New Brunswick)
2. Gather feedback regarding the intervention from cancer survivors and healthcare providers.

Participants will have access to the intervention for a period of six months. Questionnaires will be distributed to participants through the intervention at baseline, 90 days, and 180 days to assess user experience. Semi-structured interviews will be conducted with select survivor participants and healthcare providers (oncology and primary care) to determine the feasibility and acceptability of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years, capable of providing informed consent
* Diagnosed with stage I-III breast or colorectal cancer, and have completed primary treatment for their cancer (surgery and/or adjuvant systemic or radiation therapy) 6 months - 5 years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment | During enrollment
  Case report forms will be used to track recruitment metrics. The following demographics will be collected to monitor the diversity of those participating: cancer type (breast, colorectal), stage at diagnosis (in situ, stage 1, stage 2, stage 3, do not know), age (in years, prefer not to say), sex assigned at birth (male, female, intersex, prefer not to say), gender (man, woman, non-binary, other, prefer not to say), residence (rural, suburban, urban, prefer not to say), and highest level of education achieved (less than high school, high school, some post-secondary (college or university), diploma or degree, prefer not to say).
Retention | Enrollment to day 180
  Case report forms will be used to track retention metrics.
Usage of the Intervention | Baseline to day 180
  Usage metrics will be collected using the SeamlessMD software to determine the following: 1) how often the intervention was accessed by participants, 2) what elements of the intervention were accessed most, and 3) what elements of the program were utilized the least.
Survivor and Provider Acceptability and Experience | Interviews with survivor participants will be conducted after having access to the intervention for 180 days.
  Assessed via one-on-one semi-structured interviews with a sub-sample of study participants and providers at both study sites. Semi-structured interviews were chosen over focus groups for this component because the research team is seeking individual experiences with the intervention. Interviews will be carried out by a member of the research team on video conferencing software using a predetermined interview guide and will take approximately 45 minutes. The questions will center around the study participant's follow-up care experience while being supported by the intervention. Interviews with providers will focus on the feasibility and acceptability of the supportive self-management tool.

SECONDARY OUTCOMES:
Fear of Recurrence | Outcomes will be captured at baseline (study entry), on days 90 and 180, directly through the Seamless MD app software.
  Will be assessed using the 6-item Cancer Worry Scale, a validated patient-reported instrument. Cancer Worry Scale (CWS) scores range from 6 to 24 points. A score of 6 points indicates low worry, while a score of 24 points indicates very high worry.
Patient Activation | Outcomes will be captured at baseline (study entry), on days 90 and 180, directly through the Seamless MD app software.
  Will be assessed with the 13-item Patient Activation Measure (PAM), a validated patient-reported instrument. PAM includes 13 questions that produce a score on a 0-100 scale, which correlates with 1 of 4 activation levels. A level 1 score indicates low activation, while a level 4 score indicates a high activation.
Information Provision | Outcomes will be captured at baseline (study entry), on days 90 and 180, directly through the Seamless MD app software.
  There are no validated instruments to assess information provision on its own. Therefore, these will be assessed using modified survey items from the Canadian Transitions Survey, a national survey on survivors' needs and experiences after completing cancer treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Centre for Clinical Research QEII Health Sciences Centre, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No